CLINICAL TRIAL: NCT04189809
Title: Management of Hepatocellular Carcinoma : Discrepancies Between BCLC Classification and Clinical Practice in a Large Regional Multicentric Cohort
Brief Title: Discrepancies in Management of Hepatocellualr Carcinoma Between Practice and Recommendations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0572
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Chronic liver diseases; Interventional Radiology; Surgical; Therapy; resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The complex management of hepatocellular carcinoma has prompted many learned societies to issue their management recommendations or decision-making algorithms to best assist in the therapeutic decision-making of patients with HCC. Over time, the use of the BCLC algorithm (for Barcelona Clinic Liver Cancer) has become essential, at least in the West, thanks to a relatively simple and applicable classification system, and the clinical validation of numerous studies. The BCLC algorithm thus relies on the general condition of the patient, the CHILD-PUGH score reflecting hepatic function, and the tumor extension to propose one or more therapeutic solutions according to the level of scientific evidence, associating with each one. subgroups the expected survival.

While this BCLC classification has the merit of having the protocol for the management of HCC, thus avoiding many drifts related to possible local preferences, it also has many defects. For example, this classification is only rarely updated, which limits the integration of innovative therapies. Then, its design and updates were supported by the recommendations of a limited group of experts that is not necessarily representative of all the key players present daily in the management of CHC. Finally, some studies have begun to point out that this classification was interesting from a theoretical point of view, but that in practice the diversity of complex situations meant that its care recommendations were not applicable in a significant number of cases.

The objective of our study is to analyze the applicability of the BCLC classification in real-life situations. To overcome possible "center effects", the investigators analyzed in an exhaustive way the therapeutic decisions taken during the multi-disciplinary consultation meetings of 2018 and 2019 at the level of a large French region, by relying on the regional network of OncoOccitanie Oncology Record. In a second step, the investigators will analyze the causes of the discrepancies to finally propose an improvement of this BCLC classification.

ELIGIBILITY:
Inclusion criteria:

- Any patient presented at a multidisciplinary meeting within the OncoOccitanie network during the years 2018 and 2019 for the management of hepatocellular carcinoma

Exclusion criteria:

* Histological type other than CHC
* Multidisciplinary meeting that does not lead to a therapeutic decision (such as the continuation of further investigations, biopsy sampling, or active surveillance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with diagnosis of HCC proven based on tumor sampling or imaging findings
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Rate of therapeutic proposals correctly predicted by the BCLC international classification | 1 day
  Rate of therapeutic proposals correctly predicted by the BCLC international classification

SECONDARY OUTCOMES:
Rates and causes of discrepancies | 1 day
  Rates and causes of discrepancies

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC